CLINICAL TRIAL: NCT02617446
Title: The Clinical Study of the Safety and Efficacy of Istaroxime in Treatment of Acute Decompensated Heart Failure - A Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel Group Clinical Study
Brief Title: The Clinical Study of the Safety and Efficacy of Istaroxime in Treatment of Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-CV-002; 2013-000540-26 (EudraCT Number); 2015L00219 (Other: National Medical Products Administration (China))
Record Dates: First submitted 2015-07-09; First posted 2015-12-01 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: safety; efficacy; istaroxime
MeSH Terms: interventions — Istaroxime

STUDY DESIGN:
Intervention Model Description: Cohort I: Participants enrolled in a 2:1 ratio to istaroxime 0.5 µg/kg/min or placebo.
  Cohort II: Participants enrolled in a 2:1 ratio to istaroxime 1.0 µg/kg/min or placebo.
  Cohort I was enrolled first, followed by Cohort II.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): IV infusion of placebo for 24 hours
  Interventions: Drug: Placebo
- Istaroxime 0.5 µg/kg/min (Experimental): The istaroxime treatment dosed at 0.5 µg/kg/min via IV infusion for 24 hours
  Interventions: Drug: Istaroxime
- Istaroxime 1.0 µg/kg/min (Experimental): The istaroxime treatment dosed at 1.0 µg/kg/min via IV infusion for 24 hours
  Interventions: Drug: Istaroxime

INTERVENTIONS:
Drug: Placebo — IV of matching saline solution
  Arms: Placebo
Drug: Istaroxime — IV infusion of 0.5 µg/kg/min or 1.0 µg/kg/min istaroxime
  Arms: Istaroxime 0.5 µg/kg/min; Istaroxime 1.0 µg/kg/min

SUMMARY:
To assess the safety, tolerability and efficacy of two different doses of istaroxime, a new agent with lusitropic and inotropic activities that improves the cardiac contraction-relaxation cycle. The 2 doses of istaroxime (0.5 and 1.0 µg/kg/min) will be infused via i. v. for 24 hours in comparison with placebo, in treatment of Chinese and Italian patients with Acute Decompensated Heart Failure.

DETAILED DESCRIPTION:
To assess the safety, tolerability and efficacy of two different doses of istaroxime (0.5 and 1.0 µg/kg/min) in comparison with placebo, including cardiovascular and renal tolerability, as well as changes in biological markers such as N-terminal prohormone brain natriuretic peptide (NT-proBNP) and troponin T (cTnT). The study will be conducted in 96 Chinese and Italian patients with Acute Decompensated Heart Failure. This is a phase II, multicenter, randomized, double-blind, placebo-controlled, parallel group study. Patients were randomly assigned to one of two doses of istaroxime or placebo in a 2:1 ratio within two sequential cohorts of 60 patients each. This 31-day study includes a screening period (Days -1), a treatment period (Day 1), a post-treatment period (Days 2-4), and a follow-up period (which includes one patient visit on Day 30).

In all the Italian patients and in a subset of Chinese patients pharmacokinetics and metabolism of istaroxime shall also be studied.

ELIGIBILITY:
Inclusion Criteria:

Patients who fulfill the following inclusion criteria at screening will be considered for the study:

1. Signed informed consent;
2. Male or female patients 18-85 years (inclusive);
3. Admission for a recurrent acute decompensated heart failure (ADHF) episode with dyspnea at rest or minimal exertion and need of intravenous diuretic therapy (≥40 mg iv. furosemide);
4. Systolic blood pressure between 90 and 125 mmHg (limits included) without signs or symptoms of hypoperfusion including cardiogenic shock, cold extremities and peripheral vasoconstriction, oliguria/anuria, signs of cerebral hypo perfusion such as confusion;
5. Left ventricular (LV) Ejection fraction (EF) ≤ 40 % measured by 2D-Echocardiography
6. E/Ea ratio >10
7. BNP ≥ 350pg/mL or NT-pro-BNP ≥1400 pg/mL
8. Adequate echocardiography window (defined as visualization of at least 13/16 segment of the left ventricle);

Exclusion Criteria:

Any of the following criteria established at screening would render a patient ineligible for the study:

1. Pregnant or breast-feeding women (women of child bearing potential must have the results of a negative pregnancy test recorded prior to study drug administration)
2. Current (within 12 hours prior to screening) or planned (through the completion of study drug infusion) treatment with any iv. therapies, including vasodilators (including nitrates or nesiritide), positive inotropic agents and vasopressors
3. Current or need of mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device),
4. Ongoing treatment with oral digoxin. Patient treated with digoxin within the last week, can be randomised if the plasma concentration of digoxin is tested before randomization and its value will be less than 0.5 ng/ml.
5. History of hypersensitivity to the study medication or any related medication
6. Diagnosis of cardiogenic shock within the past month;
7. Acute coronary syndrome or stroke within the past 3 months;
8. Coronary artery bypass graft or percutaneous coronary intervention within the past month or planned in the next month;
9. Primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease;
10. Cor pulmonale or other causes of right-sided heart failure (HF) not related to left ventricular dysfunction;
11. Pericardial constriction or active pericarditis;
12. Atrial fibrillation with marked irregularities of heart rhythm;
13. Life threatening ventricular arrhythmia or implantable cardioverter-defibrillator (ICD) shock within the past month;
14. Cardiac resynchronization therapy (CRT), ICD, or pacemaker implantation within the past month;
15. Valvular disease as primary cause of HF;
16. Heart rate >120 bpm or < 50 bpm
17. Acute respiratory distress syndrome or ongoing sepsis;
18. Fever >38°
19. History of bronchial asthma or porphyria;
20. Donation or loss of blood equal to or exceeding 500 mL, during the 8 weeks before administration of study medication;
21. Positive testing for HIV, Hepatitis B and/or Hepatitis C;
22. Participation in another interventional study within the past 30 days;
23. The following laboratory exclusion criteria, verified based on results obtained within the last 24 hours of hospitalization:

    1. Serum creatinine > 3.0 mg/dl (> 265 µmol/L);
    2. Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) > 3 x upper limit of normal,
    3. Hemoglobin (Hb) < 10 g/dL,
    4. Platelet count < 100,000/µL,
    5. Serum potassium > 5.3 mmol/L or < 3.8 mmol/L,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2018-08-14 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Bianchi, MD, Principal Investigator — Windtree Therapeutics, Inc.
Locations (11):
- China (9):
  - Lanzhou University No.2 Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - The General Hospital Of Shenyang Military Region, Shenyang, Liaoning
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing
  - Beijing Chao Yang Hospital, Beijing
  - The 307th Hospital of Chinese People's Liberation Army, Beijing
- Italy (2):
  - University and Civil Hospital of Brescia, Brescia
  - University of Milano-Bicocca, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carubelli V, Zhang Y, Metra M, Lombardi C, Felker GM, Filippatos G, O'Connor CM, Teerlink JR, Simmons P, Segal R, Malfatto G, La Rovere MT, Li D, Han X, Yuan Z, Yao Y, Li B, Lau LF, Bianchi G, Zhang J; Istaroxime ADHF Trial Group. Treatment with 24 hour istaroxime infusion in patients hospitalised for acute heart failure: a randomised, placebo-controlled trial. Eur J Heart Fail. 2020 Sep;22(9):1684-1693. doi: 10.1002/ejhf.1743. Epub 2020 Jan 23. PMID 31975496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening to assess whether the patient qualified for the study. 144 patients were screened, 22 were determined to be screen failures and additional 2 patients were excluded for not meeting inclusion/exclusion criteria.
Groups:
- Placebo: IV infusion for 24 hours
  Placebo: IV of matching saline solution
- Istaroxime 0.5 µg/kg/Min: Istaroxime via IV infusion for 24 hours
  Istaroxime: IV infusion of istaroxime 0.5 µg/kg/min
- Istaroxime 1.0 µg/kg/Min: Istaroxime via IV infusion for 24 hours
  Istaroxime: IV infusion of istaroxime 1.0 µg/kg/min
Period: Overall Study
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Started | 39 | 41 | 40
Completed | 35 | 39 | 33
Not Completed | 4 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 5
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Death | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min | Total
Number analyzed (Participants) | 39 | 41 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.67 (16.21) | 59.73 (15.53) | 52.23 (13.02) | 56.24 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 18
  Male | 34 | 34 | 34 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 32 | 24 | 40 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 17 | 0 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 32 | 24 | 40 | 96
  Italy | 7 | 17 | 0 | 24
E/Ea Ratio [Mean (Standard Deviation); unit: Unitless ratio] — Unitless ratio of E (cm/sec) to Ea (cm/sec) as measured by echocardiogram. The endpoint is the Tissue Doppler echocardiography showing measurement of mitral E/e' ratio for assessment of diastolic dysfunction. Initially mitral E wave is measured. After that, color Tissue Doppler (tissue velocity imaging or TVI) mode is switched on to assess tissue Doppler. The cursor is placed over the medial mitral annulus and tissue Doppler tracing obtained. This allows e' velocity to be measured. Higher values are suggestive of a worse outcome; less than 8 is normal. Population: Measurements for 1 istaroxime 0.5 µg/kg/min participant not recorded (missing).
  Unitless ratio
    number analyzed (Participants) | 39 | 40 | 40 | 119
    (all) | 17.0 (5.33) | 20.4 (7.87) | 15.1 (5.48) | 17.5 (6.36)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: % of blood in heart pumped] — LVEF (% blood ejected from heart) as measured by echocardiogram Population: Measurements for 4 participants (1 placebo participant, 1 istaroxime 0.5 µg/kg/min participant, 2 istaroxime 1.0 µg/kg/min participants) not recorded (missing)
  % of blood in heart pumped
    number analyzed (Participants) | 38 | 40 | 38 | 116
    (all) | 26.2 (7.4) | 27.4 (6.7) | 28.7 (7.2) | 27.4 (7.1)
Stroke Volume Index [Mean (Standard Deviation); unit: ml/m²] — Stroke volume index (SVI) as measured by echocardiogram Population: Measurements for 2 participants (1 istaroxime 0.5 µg/kg/min participant, 1 istaroxime 1.0 µg/kg/min participant) not recorded (missing)
  ml/m²
    number analyzed (Participants) | 39 | 40 | 39 | 118
    (all) | 21.6 (7.73) | 25.9 (7.10) | 17.1 (5.69) | 21.6 (6.89)
Dyspnea [Mean (Standard Deviation); unit: Scores on a scale] — Scores on a scale using Visual Analog Scales (VAS). Scores range from 0 to 100, with higher values indicating a better outcome (less dyspnea).
  Scores on a scale | 70.8 (21.32) | 73.6 (19.49) | 71.5 (20.95) | 72.0 (20.59)
Troponin (cTnT) [Mean (Standard Deviation); unit: ng/L] — Cardiac muscle troponin T (cTnT) measured as ng/L
  ng/L | 33.5 (33.9) | 34.2 (36.6) | 40.4 (78.3) | 36.0 (53.6)
eGFR [Mean (Standard Deviation); unit: ml/min/1.73·m²] — Estimated glomerular filtration rate (eGFR), measured as ml/min/1.73·m² Population: Measurements for 1 istaroxime 0.5 µg/kg/min participant not recorded (missing)
  ml/min/1.73·m²
    number analyzed (Participants) | 39 | 40 | 40 | 119
    (all) | 78.1 (38.33) | 72.3 (30.93) | 81.3 (27.01) | 77.2 (32.36)

OUTCOME MEASURES:

1. Primary Outcome: Change in E/Ea Ratio
Description: Change from baseline at 24 hours in the unitless ratio of E (cm/sec) to Ea (or e') (cm/sec) as measured by echocardiogram.
  The endpoint is the Tissue Doppler echocardiography showing measurement of mitral E/Ea ratio for assessment of diastolic dysfunction. Initially mitral E wave is measured. After that, color Tissue Doppler (tissue velocity imaging or TVI) mode is switched on to assess tissue Doppler. The cursor is placed over the medial mitral annulus and tissue Doppler tracing obtained. This allows Ea velocity to be measured. Higher values are suggestive of a worse outcome; less than 8 is normal.
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless ratio
Groups:
- Istaroxime 0.5 µg/kg/Min: Istaroxime participants receiving 0.5 µg/kg/min (Cohort I)
- Placebo Cohort I: Placebo participants enrolled in Cohort I
- Istaroxime 1.0 µg/kg/Min: Istaroxime participants receiving 1.0 µg/kg/min (Cohort II)
- Placebo Cohort II: Placebo participants enrolled in Cohort II
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
Unitless ratio | -4.55 [-6.05 to -3.04] | -1.55 [-3.77 to 0.67] | -3.16 [-4.09 to -2.24] | -1.08 [-2.30 to 0.13]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in E/Ea ratio between istaroxime and placebo; Test type: Superiority; p = 0.029, ANOVA — Alpha set at 0.05; Treatment term included in the model; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-5.68 to -0.32]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in E/Ea ratio between istaroxime and placebo; Test type: Superiority; p = 0.009, ANOVA — Alpha set at 0.05; Treatment term included in the model; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-3.61 to -0.55]

2. Secondary Outcome: Change in LVEF
Description: Change from baseline at 24 hours in LV ejection fraction (LVEF) by tissue Doppler
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Mean (95% Confidence Interval); unit: % of blood leaving the heart
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
% of blood leaving the heart | 3.026 [1.850 to 4.203] | 1.263 [-0.401 to 2.927] | 3.818 [2.362 to 5.275] | 2.833 [0.861 to 4.805]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in LVEF % between istaroxime and placebo participants; Test type: Superiority; p = 0.089, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term included in the model; Mean Difference (Final Values) = 1.7632, 95% CI 2-sided [-0.2751 to 3.8014]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in LVEF % between istaroxime and placebo participants; Test type: Superiority; p = 0.423, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term included in the model; Mean Difference (Final Values) = 0.9848, 95% CI 2-sided [-1.4668 to 3.4365]

3. Secondary Outcome: Change in SVI
Description: Change from baseline at 24 hours in stroke volume index (SVI) by tissue Doppler
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/m²
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
mL/m² | 5.334 [3.371 to 7.296] | 1.649 [-1.126 to 4.425] | 5.488 [3.882 to 7.094] | 3.178 [1.030 to 5.327]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in SVI between istaroxime and placebo participants; Test type: Superiority; p = 0.034, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = 3.684, 95% CI 2-sided [0.285 to 7.083]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in E to A ratio between istaroxime and placebo participants; Test type: Superiority; p = 0.090, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = 2.310, 95% CI 2-sided [-0.373 to 4.992]

4. Secondary Outcome: Change in E/A Ratio
Description: Change from baseline at 24 hours in E/A ratio by tissue Doppler
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless ratio
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
Unitless ratio | -0.643 [-1.091 to -0.197] | 0.133 [-0.463 to 0.729] | -0.654 [-1.093 to -0.216] | 0.175 [-0.419 to 0.769]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in E to A ratio between istaroxime and placebo participants; Test type: Superiority; p = 0.042, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is included in the model; Mean Difference (Final Values) = -0.777, 95% CI 2-sided [-1.522 to -0.032]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in E to A ratio between istaroxime and placebo participants; Test type: Superiority; p = 0.029, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = -0.829, 95% CI 2-sided [-1.568 to -0.091]

5. Secondary Outcome: Change in LV End Systolic Volume
Description: Change from baseline in left ventricular end systolic volume (LVESV) by tissue Doppler
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
mL | -7.105 [-10.933 to -3.277] | -1.736 [-7.150 to 3.677] | -11.39 [-17.438 to -5.350] | -11.83 [-20.017 to -3.649]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in LVESV between istaroxime and placebo participants; Test type: Superiority; p = 0.110, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = -5.368, 95% CI 2-sided [-11.999 to 1.262]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in LVEDV between istaroxime and placebo participants; Test type: Superiority; p = 0.931, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = 0.439, 95% CI 2-sided [-9.735 to 10.614]

6. Secondary Outcome: Change in LV End Diastolic Volume
Description: Change from baseline in left ventricular end diastolic volume (LVEDV) by tissue Doppler
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Istaroxime 0.5 µg/kg/Min | Placebo Cohort I | Istaroxime 1.0 µg/kg/Min | Placebo Cohort II
Number analyzed (Participants) | 41 | 19 | 40 | 20
mL | -0.710 [-4.243 to 2.822] | 0.947 [-4.049 to 5.944] | -3.666 [-9.507 to 2.173] | -7.611 [-15.518 to 0.296]
Statistical Analysis 1: Comparison: Istaroxime 0.5 µg/kg/Min vs Placebo Cohort I; Null hypothesis: No difference in E to A ratio between istaroxime and placebo participants; Test type: Superiority; p = 0.589, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term in the model; Mean Difference (Final Values) = -1.657, 95% CI 2-sided [-7.777 to 4.461]
Statistical Analysis 2: Comparison: Istaroxime 1.0 µg/kg/Min vs Placebo Cohort II; Null hypothesis: No difference in E to A ratio between istaroxime and placebo participants; Test type: Superiority; p = 0.424, ANOVA — Alpha set at 0.05. No adjustment for multiple comparisons; Treatment term is in the model; Mean Difference (Final Values) = 3.944, 95% CI 2-sided [-5.886 to 13.774]

7. Secondary Outcome: Change in Dyspnea
Description: Measured using a visual analog scale (0 to 100). Higher scores indicate less dyspnea.
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Score on a scale (Visual Analog Scale)
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Score on a scale (Visual Analog Scale) | 9.75 (11.80) | 9.14 (10.08) | 12.09 (14.79)
Statistical Analysis 1: Comparison: Placebo vs Istaroxime 0.5 µg/kg/Min; Null hypothesis: no difference between treatment groups; Test type: Superiority — Linear mixed model with treatment, center, timepoint, gender, baseline cTnT value, atrial fibrillation, and treatment*timepoint interaction included in the model; p = 0.987, Mixed Models Analysis — Unadjusted alpha of 0.05 is the threshold for statistical significance; Kenward-Roger adjustment used for the degrees of freedom; Mean Difference (Final Values) = -0.041, 95% CI 2-sided [-5.216 to 5.133]
Statistical Analysis 2: Comparison: Placebo vs Istaroxime 1.0 µg/kg/Min; Null hypothesis: no difference between treatment groups; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.251, Mixed Models Analysis — Unadjusted alpha of 0.05 is the threshold for statistical significance; Kenward-Roger adjustment used for the degrees of freedom; Mean Difference (Final Values) = 3.015, 95% CI 2-sided [-2.168 to 8.198]

8. Other Pre Specified Outcome: Change in cTnT
Description: Safety endpoint: Changes in troponin (cTnT)
Time Frame: 24 hours
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
ng/L | 0.23 (10.83) | 0.51 (7.58) | -4.06 (49.97)

9. Other Pre Specified Outcome: Change in eGFR
Description: Safety endpoint: Change from baseline in estimated glomerular filtration rate (eGFR)
Time Frame: 24 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ml/min/1.73·m²
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
ml/min/1.73·m² | -0.60 (14.71) | 5.19 (16.25) | 7.65 (13.22)

10. Other Pre Specified Outcome: Participants With Clinically or Hemodynamically Significant Episodes of Arrhythmias
Description: Safety endpoint: Number of participants with incidence of clinically or hemodynamically significant episodes of supraventricular or ventricular arrhythmias detected by continuous ECG dynamic monitoring
Time Frame: 24 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants | 6 | 1 | 4

11. Other Pre Specified Outcome: PR Interval
Description: Safety Endpoint: The PR interval, measured in milliseconds, extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex (the onset of ventricular depolarization).
Time Frame: 24 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
msec | 184.0 (31.27) | 179.2 (28.11) | 169.41 (32.72)

12. Other Pre Specified Outcome: QRS Duration
Description: Safety endpoint: The quasi-random signal (QRS) duration represents the time for ventricular depolarization, normally 0.06 to 0.10 seconds.
Time Frame: 24 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
msec | 125.2 (37.11) | 132.5 (31.59) | 127.6 (26.65)

13. Other Pre Specified Outcome: QTc Interval
Description: Safety Endpoint: The corrected QT interval (QTc) on an ECG represents the duration in milliseconds of the ventricular action potential, which physiologically correlates with the duration of the ventricular depolarization and repolarization.
Time Frame: 24 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
msec | 472.8 (41.90) | 480.8 (55.72) | 486.9 (40.18)

14. Other Pre Specified Outcome: All-Cause Mortality at Day 30
Description: Safety endpoint: Mortality at Day 30
Time Frame: 30 days
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants | 0 | 0 | 2

15. Other Pre Specified Outcome: RBC - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in red blood cells (RBC)
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 22 | 17 | 21
  Normal to Abnormal | 5 | 3 | 4
  Abnormal to Normal | 2 | 3 | 4
  Abnormal to Abnormal | 8 | 16 | 7
  Missing | 2 | 2 | 4

16. Other Pre Specified Outcome: Hematocrit - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in hematocrit
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 21 | 15 | 17
  Normal to Abnormal | 7 | 3 | 5
  Abnormal to Normal | 3 | 7 | 6
  Abnormal to Abnormal | 6 | 14 | 8
  Missing | 2 | 2 | 4

17. Other Pre Specified Outcome: Hemoglobin - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in hemoglobin
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 23 | 13 | 23
  Normal to Abnormal | 5 | 3 | 2
  Abnormal to Normal | 1 | 7 | 5
  Abnormal to Abnormal | 8 | 16 | 6
  Missing | 2 | 2 | 4

18. Other Pre Specified Outcome: White Blood Cells (WBC) - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in WBC
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 35 | 30 | 25
  Normal to Abnormal | 2 | 6 | 6
  Abnormal to Normal | 0 | 1 | 2
  Abnormal to Abnormal | 0 | 2 | 3
  Missing | 2 | 2 | 4

19. Other Pre Specified Outcome: Platelets - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in platelets
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 26 | 32 | 31
  Normal to Abnormal | 3 | 2 | 4
  Abnormal to Normal | 4 | 1 | 0
  Abnormal to Abnormal | 4 | 3 | 1
  Missing | 2 | 3 | 4

20. Other Pre Specified Outcome: Potassium - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in potassium
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 37 | 40 | 34
  Normal to Abnormal | 1 | 0 | 2
  Abnormal to Normal | 0 | 0 | 0
  Abnormal to Abnormal | 0 | 0 | 0
  Missing | 1 | 1 | 4

21. Other Pre Specified Outcome: Sodium - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in sodium
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 23 | 21 | 19
  Normal to Abnormal | 9 | 12 | 8
  Abnormal to Normal | 4 | 2 | 1
  Abnormal to Abnormal | 2 | 5 | 8
  Missing | 1 | 1 | 4

22. Other Pre Specified Outcome: Calcium - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in calcium
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 24 | 26 | 20
  Normal to Abnormal | 4 | 2 | 1
  Abnormal to Normal | 3 | 2 | 9
  Abnormal to Abnormal | 3 | 1 | 4
  Missing | 5 | 10 | 6

23. Other Pre Specified Outcome: BUN - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in blood urea nitrogen (BUN)
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 11 | 13 | 14
  Normal to Abnormal | 7 | 4 | 6
  Abnormal to Normal | 3 | 2 | 8
  Abnormal to Abnormal | 14 | 16 | 7
  Missing | 4 | 6 | 5

24. Other Pre Specified Outcome: ALT - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in alanine aminotransferase (ALT)
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 29 | 31 | 29
  Normal to Abnormal | 1 | 1 | 2
  Abnormal to Normal | 2 | 1 | 0
  Abnormal to Abnormal | 4 | 5 | 5
  Missing | 3 | 3 | 4

25. Other Pre Specified Outcome: AST - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in aspartate aminotransferase (AST)
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 28 | 28 | 24
  Normal to Abnormal | 1 | 4 | 5
  Abnormal to Normal | 3 | 1 | 4
  Abnormal to Abnormal | 4 | 4 | 3
  Missing | 3 | 4 | 4

26. Other Pre Specified Outcome: Total Bilirubin - Shift
Description: Safety endpoint: Baseline normal/abnormal to Day 3 normal/abnormal in total bilirubin
Time Frame: Day 3
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
Number analyzed (Participants) | 39 | 41 | 40
Participants
  Normal to Normal | 9 | 21 | 13
  Normal to Abnormal | 3 | 2 | 2
  Abnormal to Normal | 9 | 3 | 6
  Abnormal to Abnormal | 13 | 11 | 15
  Missing | 5 | 4 | 4

ADVERSE EVENTS:
Time Frame: Enrollment to 30 days after enrollment
Description: Participants were closely supervised in a hospital. Adverse events were observed by study staff and reported by participants.
Arm/Group | Placebo | Istaroxime 0.5 µg/kg/Min | Istaroxime 1.0 µg/kg/Min
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 2/40
Serious Adverse Events (participants affected / at risk) | 2/39 | 2/41 | 6/40
Other Adverse Events (participants affected / at risk) | 23/39 | 31/41 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Istaroxime 0.5 µg/kg/Min (N=41) | Istaroxime 1.0 µg/kg/Min (N=40)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal embolism (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Istaroxime 0.5 µg/kg/Min (N=41) | Istaroxime 1.0 µg/kg/Min (N=40)
Arrythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (4) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 9 (10)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 10 (10)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 2 (3) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 17 (17) | 12 (12) — Includes "Implant site pain", "Infusion site pain", and "Injection site pain"
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood urea increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Blood uric acid increased (Investigations) | 3 (3) | 3 (3) | 2 (2)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 3 (3) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
The major limitation of this study regards enrollment discrepancies between the study populations and sites of the two cohorts, with Cohort 2 enrolling exclusively Asian patients. We observed that patients enrolled in this trial were younger and with a better renal function compared to other studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data and results of the clinical study are possessed by sponsor and investigator. Investigator agrees not to submit the results of this study for publication or presentation before the sponsor review the accuracy and no leakage of confidential information in the manuscript.

DOCUMENTS (3):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT02617446/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT02617446/SAP_001.pdf
  • Informed Consent Form (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02617446/ICF_002.pdf